CLINICAL TRIAL: NCT07380711
Title: Prospective and Retrospective Observational Real-world Study to Characterize Patients With COPD on Dupilumab Long-term Treatment, and Assess Safety and Patient Reported Outcomes
Brief Title: Long-term Real-world Study of Dupilumab in COPD : Patient Characteristics, Safety and Patient-reported Outcomes
Acronym: AURORA
Status: Recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS19236
Record Dates: First submitted 2026-01-13; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Chronic Obstructive Pulmonary Disease COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

GROUPS / COHORTS (1):
- Treated cohort: Dupilumab

SUMMARY:
The OBS19236 is a retrospective and prospective, non-interventional observational study in COPD patients treated with dupilumab as part of routine clinical care. It will follow-up about 350 to 500 participants over 36 months in up to 50 sites in France.

DETAILED DESCRIPTION:
Study duration per participant is expected to be approximately 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing and able to sign informed consent for use of their pseudonymized clinical data within the present non-intervention study.
* Adult patients.
* Patients with uncontrolled Chronic Obstructive Pulmonary Disease (COPD) despite long-acting muscarinic antagonist (LAMA)/ Long-acting beta2-agonist (LABA)/ Inhaled Corticosteroid (ICS) (or LAMA/LABA if ICS are not appropriate) therapy and elevated blood eosinophils (a blood eosinophil count ≥ 300 cells/microL).
* Patients newly initiated on dupilumab treatment as indicated in the dupilumab summary of product characteristics (SmPC) in the specified label for COPD, determined by the treating physician, and independent of participation in the non-interventional study (NIS).

Exclusion Criteria:

* Patient not eligible for dupilumab treatment according to SmPC.
* Participation in an ongoing interventional study or participation in an interventional study up to 12 months before enrolment that might, in the treating physician's opinion, influence the assessments for the current study.
* Any acute or chronic condition that, in the treating physician´s opinion, would limit the patient´s ability to complete questionnaires or to participate in this study or impact the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is planned to recruit 350 to 500 participants, in up to 50 sites in France.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2030-08-14 (Estimated); Study Completion 2030-08-14 (Estimated)

PRIMARY OUTCOMES:
Descriptive statistical analysis of socio-demographics | Baseline
Descriptive statistical analysis of medical disease | Baseline
Descriptive statistical analysis of treatment history | Baseline
Descriptive statistical analysis of clinical disease characteristics (symptoms) | In the 1 year prior to Dupilumab initiation
Descriptive statistical analysis of clinical disease characteristics (exacerbations) | In the 2 years prior to Dupilumab initiation
Descriptive statistical analysis of clinical disease characteristics (lung function parameters) | In the 1 year prior to Dupilumab initiation
Descriptive statistical analysis of clinical disease characteristics (max eosinophils [EOS]) | In the 1 year prior to Dupilumab initiation
Descriptive statistical analysis of clinical disease characteristics (fractional exhaled nitric oxide [FeNO] levels) | In the 1 year prior to Dupilumab initiation
Descriptive statistical analysis of clinical disease characteristics (immunoglobulin E [IgE] levels) | In the 1 year prior to Dupilumab initiation
Descriptive statistical analysis of clinical disease characteristics (Global Initiative for Chronic Obstructive Lung Disease (GOLD) grade and group) | Baseline
Descriptive statistical analysis of clinical disease characteristics (smoking status and pack years (tobacco and cannabis)) | Baseline
Descriptive statistical analysis of clinical disease characteristics (treated asthma in childhood and concomitant asthma according to the investigator opinion,) | Baseline
Descriptive statistical analysis of clinical disease characteristics (Cardiovascular (CV)) comorbidities) | Baseline
Descriptive statistical analysis of clinical disease characteristics (Otorhinolaryngology (ORL) comorbidities) | Baseline
Descriptive statistical analysis of clinical disease characteristics (date of Chronic Obstructive Pulmonary Disease (COPD) diagnosis) | Baseline
Date of COPD diagnosis and GOLD grade/group at COPD diagnosis | Baseline
Descriptive statistical analysis of clinical disease characteristics (BODE and/or BODEx scores-index for COPD survival) | Baseline
Descriptive statistical analysis of clinical disease characteristics (history of pulmonary rehabilitation) | Baseline
Descriptive statistical analysis of Hospital Anxiety and Depression scale (HADS). | Baseline
  Score range 0-42, higher values indicating a worse outcome
Descriptive statistical analysis of Vaccine status. | Baseline
Descriptive statistical analysis of Emphysema assessment according to treating physician, based on CT scan | In the last 3 years prior to treatment initiation

SECONDARY OUTCOMES:
Annualized rate of Chronic Obstructive Pulmonary Disease (COPD) exacerbations | After 12, 24 and 36 months compared to the year before baseline.
Change in exacerbation rate | From treatment start to month 6, 12, 24 and 36.
Time to first exacerbation | Since Dupilumab initiation and during the study period (3 years)
Cumulative moderate and severe exacerbations | Since Dupilumab initiation and during the study period (3 years)
Change over time in pre- and post-bronchodilator forced expiratory volume in 1 second (FEV1) | From treatment start to month 6, 12, 24 and 36.
Change over time in pre- and post-bronchodilator Forced Vital Capacity (FVC) | From treatment start to month 6, 12, 24 and 36
Change over time in pre- and post- bronchodilator forced expiratory volume in 1 second (FEV1)/ Forced vital capacity (FVC) | From treatment start to month 6, 12, 24 and 36
Change over time in COPD Assessment Test (CAT) Score | From treatment start to month 6, 12, 24 and 36.
  Score range 0-40, higher values indicating a worse outcome
Change over time in modified Medical Research Council (mMRC) score | From treatment start to month 6, 12, 24 and 36.
  Score range 0-4, higher values indicating a worse outcome
Number of hospitalizations during dupilumab treatment vs. the year before dupilumab initiation | After 6, 12, 24 and 36 months of dupilumab treatment vs. the year before dupilumab initiation
Reason(s) for discontinuation of dupilumab treatment | Month 6, 12, 24, and 36
Frequency and type of Adverse events (AEs) | During the study period (3 years)
Frequency and type of possible dupilumab-related treatment-emergent adverse events (TEAEs) | During the study period (3 years)

OTHER OUTCOMES:
Change over time in the Residual Volume (RV) | From treatment start to months 6, 12, 24 and 36.
Change over time in the Functional Residual Capacity (FRC) | From treatment start to months 6, 12, 24 and 36.
Change over time in the Diffusion Lung Capacity for Carbon Monoxide [DLCO] | From treatment start to months 6, 12, 24 and 36.
Number of missed workdays due to Chronic Obstructive Pulmonary Disease (COPD) | After 6, 12, 24 and 36 months of dupilumab treatment vs. the year before baseline
Number of major adverse cardiovascular events (MACE) | After 6, 12, 24 and 36 months of dupilumab treatment vs. the year before baseline

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Investigational Site Number : 2500034, Pierre-Bénite
  - Investigational Site Number : 2500035, Villeurbanne

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org